CLINICAL TRIAL: NCT00168740
Title: Pivotal Phase III Multi-Center Study to Evaluate the Safety and Efficacy of Once Weekly Times Four Dosing of IDEC-C2B8 (IDEC-102) in Patients With Relapsed Low-Grade or Follicular B-Cell Lymphoma
Brief Title: Treatment of Relapsed Low-Grade or Follicular Lymphoma With Rituximab (Also Known as Rituxan, IDEC-C2B8, IDEC-102)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDEC-102-05
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Low-Grade or Follicular B-Cell Non-Hodgkin's Lymphoma
Keywords: rituximab; Rituxan; B-cell lymphoma; low-grade; follicular; anti-CD20 monoclonal antibody
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab

INTERVENTIONS:
Drug: rituximab

SUMMARY:
Rituximab is an antibody made in a laboratory. It binds to lymphoma cells and kills them. Treatment of recurrent B-cell lymphoma with rituximab may delay or prevent relapses. A total of 166 patients with recurrent B-cell lymphoma were given intravenous rituximab once a week for 4 weeks. The patients' tumors were measured before and after treatment. Ten patients had a complete response and 70 patients had a partial response to rituximab. The median duration of response was 11.2 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed, low-grade or follicular B-cell lymphoma
* CD20-positive lymphoma
* Progressive, measurable disease
* Sign informed consent
* 3 weeks beyond standard therapy
* Good performance status
* Adequate hematologic, renal, and hepatic function

Exclusion Criteria:

* Chronic lymphocytic leukemia
* Lesions greater than or equal to 10 cm in diameter
* CNS lymphoma
* AIDS-related lymphoma
* Pleural effusions or ascites secondary to lymphoma
* Active, opportunistic infection
* Serious nonmalignant disease
* Prior investigational therapies, including prior anti-CD20 therapy
* Recent major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1995-04

PRIMARY OUTCOMES:
overall response rate

SECONDARY OUTCOMES:
time to disease progression
progressive disease-free interval

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J. Grillo-Lopez, M.D., Study Director — Biogen
Locations (31):
- United States (29):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Natioal Medical Center, Duarte, California
  - Scripps Memorial Hospital, La Jolla, California
  - UCSD Stem Cell Laboratory, La Jolla, California
  - Hoag Hospital, Newport Beach, California
  - Sutter Cancer Center, Sacramento, California
  - Sidney Kimmel Cancer Center, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Robert H. Lurie Cancer Center, Northwestern University, Chicago, Illinois
  - University of Iowa General Hospital, Iowa City, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Louisiana State University, Shreveport, Louisiana
  - University of Maryland Cancer Center, Baltimore, Maryland
  - Michigan State University, East Lansing, Michigan
  - St. Louis University Medical Center, St Louis, Missouri
  - Roswell Park Cancer Center, Buffalo, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The West Clinic, P.C., Memphis, Tennessee
  - Texas Oncology, P.A., Dallas, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Canada (2):
  - Ottawa General Hospital, Ottawa, Ontario
  - Toronto-Sunnybrook Regional Cancer Center, Toronto, Ontario

REFERENCES:
- [Result] McLaughlin P, Grillo-Lopez AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol. 1998 Aug;16(8):2825-33. doi: 10.1200/JCO.1998.16.8.2825. PMID 9704735